CLINICAL TRIAL: NCT01654302
Title: Efficacy and Safety of Synera in OA Pain
Brief Title: Efficacy and Safety of Synera in Osteoarthritis Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas J. Schnitzer (Other)
Collaborators: Nuvo Research Inc. (Industry)
Responsible Party: Sponsor-Investigator, Thomas J. Schnitzer, Professor, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00061115
Record Dates: First submitted 2012-07-11; First posted 2012-07-31 (Estimated); Results first posted 2014-11-10 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Lidocaine; Tetracaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Synera (Active Comparator): lidocaine/tetracaine patch with heating component which consists of iron powder, activated carbon, sodium chloride, wood flour, water and filter paper.
  Interventions: Drug: Synera
- Inactive Patch (Placebo Comparator): placebo patch identical in appearance and composition (namely, the heating components) to the active patch other than lacking the lidocaine and tetracaine active ingredients.
  Interventions: Drug: Inactive patch

INTERVENTIONS:
Drug: Synera — 70 mg lidocaine/ 70 mg tetracaine topical patch applied once for 12 hours
  Other Names: lidocaine/tetracaine
  Arms: Synera
Drug: Inactive patch — placebo patch applied once for 12 hours
  Other Names: placebo
  Arms: Inactive Patch

SUMMARY:
Knee osteoarthritis (OA) can result in significant pain and limitation of function. A number of topical non-steroidal anti-inflammatory drugs have been shown to reduce pain in this condition. This study examines a different topical approach, utilizing a topical anesthetic agent, to evaluate if application of such an agent would provide relief of exercise-induced knee pain in people with knee OA.

DETAILED DESCRIPTION:
Subjects participated in two visits each at least 1 week apart, where they underwent two exercise interventions - a baseline exercise without treatment and a experimental exercise with intervention (Synera patch or Inactive patch). Participants rated their pain on a NRS-11 1 minute, 5 minutes, and 60 minutes after both exercises, as well as 6 hours after the experimental exercise, before bedtime, and the following morning. Subjects were randomized to receive either Synera at the first visit and the inactive patch at the second visit or the inactive patch at the first visit and Synera patch at the second visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 40 years and above
2. Meet American College of Rheumatology criteria for knee OA
3. Knee pain most days of the week for the past month
4. Knee pain > 5/10 after exercise intervention
5. Capable of undertaking exercise intervention
6. Stable cardiovascular function
7. Able to return for all clinic visits
8. Able to read and understand the informed consent document

Exclusion Criteria:

1. Use of a walker to ambulate or inability to ambulate
2. Other forms of arthritis
3. Other major causes of pain that could be expected to interfere with assessment of pain during this trial, e.g., recurrent migraine, back pain, fibromyalgia
4. History of myocardial infarction
5. Blood Pressure > 140 systolic/100 diastolic
6. Scheduled for and likely to need joint replacement surgery in the next 3 months
7. Any medical condition that in the judgment of the investigator would make the participant not suitable for the study
8. Sensitivity to lidocaine, topical or injectable analgesics/anesthetics.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnitzer, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Synera Then Placebo: Subjects received the Synera patch during the First Intervention (Day 1) and the Inactive patch at the Second Intervention (Day 7).
- Placebo Then Synera: Subjects received the Inactive patch (placebo) during the First Intervention (Day 1) and the Synera patch at the Second Intervention (Day 7).
Period: First Intervention (Day 1)
Arm/Group | Synera Then Placebo | Placebo Then Synera
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Intervention (Day 7)
Arm/Group | Synera Then Placebo | Placebo Then Synera
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis performed for participants that completed study.
Groups:
- Synera Then Placebo: Subjects received the Synera patch during the First Intervention (Day 1) and the Inactive patch (placebo) at the Second Intervention (Day 7).
- Total: Total of all reporting groups
Arm/Group | Synera Then Placebo | Placebo Then Synera | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (7.01) | 60 (8.26) | 58 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 15 | 23
  Male | 11 | 4 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 14 | 29
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Baseline Index Knee Pain Scores [Mean (Standard Deviation); unit: units on a scale] — Subject average baseline index knee pain scores are reported prior to intervention for each group - Synera then Placebo and Placebo then Synera. Index knee pain was reported using the Numeric Rating Scale, a scale from 0 to 10 where 0 = no pain and 10 = the worst pain possible.
  units on a scale | 5.90 (1.25) | 6.26 (1.37) | 6.08 (1.33)

OUTCOME MEASURES:

1. Primary Outcome: Index Knee Pain Scores on a Numeric Rating Scale (NRS)
Description: Subject rated index knee pain 5 minutes after stopped experimental exercise (with intervention). Index knee pain was reported using the Numeric Rating Scale, a scale from 0 to 10 where 0 = no pain and 10 = the worst pain possible.
Time Frame: 5 minutes after stopped exercise, performed 1 hour after intervention (patch application)
Population: Of the 40 subjects 2 were lost to follow-up, one from each group, making a total of 38 participants included in the analysis. Unfortunately, NRS data at 5 minutes post-exercise is missing for 2 subjects in the Synera treatment group and 1 subject in the Placebo group due to technical errors. The data was captured but we were unable to retrieve it.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Synera: 70 mg lidocaine/ 70 mg tetracaine topical patch: 70 mg lidocaine/ 70 mg tetracaine topical patch applied once for 12 hours
- Inactive Patch: placebo: placebo
Arm/Group | Synera | Inactive Patch
Number analyzed (Participants) | 36 | 37
units on a scale | 4.167 (2.242) | 4.703 (2.253)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Synera | Inactive Patch
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 6/39 | 2/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synera (N=39) | Inactive Patch (N=39)
Errythmia (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No